CLINICAL TRIAL: NCT02285140
Title: Prevention of Infections in Cardiac Surgery: a Cluster-randomized Factorial Cross-over Trial
Brief Title: Prevention of Infections in Cardiac Surgery
Acronym: PICS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding received for eventual full trial, and data rolled over into full trial. Full trial registered under NCT06567808.
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Dominik Mertz, Assistant Professor, Medical Director Infection Prevention and Control, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: PICS Vanguard
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Thoracic Surgery; Antibiotic Prophylaxis
MeSH Terms: interventions — Cefazolin; Vancomycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cefazolin monotherapy, short course (Experimental): One pre-op dose of cefazolin 30-60 minutes prior to surgery followed by a second dose either four hours after the first dose or upon wound closure (whatever comes first) will be administered
  Interventions: Drug: Cefazolin
- Cefazolin monotherapy, long course (Experimental): One pre-op dose of cefazolin 30-60 minutes prior to surgery followed by a second dose either four hours after the first dose or upon wound closure (whatever comes first) will be administered followed by additional five doses every eight hours postoperatively (last dose 44 hours after the first dose).
  Interventions: Drug: Cefazolin
- Combination therapy, short course (Experimental): One pre-op dose of cefazolin 30-60 minutes prior to surgery followed by a second dose either four hours after the first dose or upon wound closure (whatever comes first) will be administered. In addition, one dose of vancomycin 60-90min pre-op will be administered.
  Interventions: Drug: Cefazolin; Drug: Vancomycin
- Combination therapy, long course (Experimental): One pre-op dose of cefazolin 30-60 minutes prior to surgery followed by a second dose either four hours after the first dose or upon wound closure (whatever comes first) will be administered followed by additional five doses every eight hours postoperatively (last dose 44 hours after the first dose). In addition, one dose of vancomycin 60-90min pre-op will be administered followed by 3 post-op doses every 12 hours (last dose 36 hours after first dose)
  Interventions: Drug: Cefazolin; Drug: Vancomycin

INTERVENTIONS:
Drug: Cefazolin — administration as outlined
Drug: Vancomycin — administration as outlined
  Arms: Combination therapy, long course; Combination therapy, short course

SUMMARY:
There is clinical equipoise about the question of whether antibiotic prophylaxis should be given for a short period or an extended period of time as reflected by inconsistencies in major guidelines, current practices at Canadian centers, and as concluded in the three systematic reviews. There also is clinical equipoise on whether the addition of vancomycin to routine cefazolin prophylaxis can further reduce s-SSI rates. A short duration of combined antimicrobial prophylaxis can reduce side effects of exposure to antimicrobials such as infections with C. difficile or emergence of resistance, but may also reduce the incidence of s-SSIs. The objective of the eventual full scale study is to determine whether adding vancomycin to cefazolin can reduce SSIs as well as whether short-term prophylaxis is as effective as long-term prophylaxis. The rationale to conduct the proposed pilot study is to assess the feasibility to conduct this factorial cluster randomized cross-over trial, the adherence to the study protocol at each pilot site, the length of time to fill out the case report forms, and to get reliable estimates of event rates for sample size calculation for the main study

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (≥18 years of age) undergoing open-heart surgery (sternotomy, including minimally-invasive surgical techniques).

Exclusion Criteria:

* Patients on antibiotics at the time of surgery.
* Previous enrollment in this trial.
* Known MRSA carriers. Beta-lactam allergy (IgE-mediated) precluding the use of cefazolin
* Participant in another study that may interfere with this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5989 (Actual)
Dates: Start 2015-04; Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients receiving antibiotics according to study protocol | 3 months post-surgery
  Co-Primary outcome of pilot study
Proportion of patients with complete follow-up, i.e. up to 90 days or death; goal >95% | 3 months post-surgery
  Co-Primary outcome of pilot study
Agreement of blinded outcome assessment based on information from the case report form | 3 months post-surgery
  Co-Primary outcome of pilot study

SECONDARY OUTCOMES:
Deep incisional and organ/space sternal surgical site infection (NHSN/CDC) | 3 months post-surgery
  Primary outcome of eventual full trial
All types of sternal surgical site infection (superficial, deep, organ; NHSN/CDC) | 3 months post-surgery
  Secondary outcome of eventual full trial
Mortality | 3 months post-surgery
  Secondary outcome of eventual full trial
Clostridium difficile infection | 3 months post-surgery
  Secondary outcome of eventual full trial

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Mertz, MD, MSc, Principal Investigator — Hamilton Health Sciences Corporation
Locations (4):
- Canada (4):
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Jewish Hospital, Montreal, Quebec
  - University of Sherbrook, Sherbrook, Quebec

REFERENCES:
- [Derived] van Oostveen RB, Romero-Palacios A, Whitlock R, Lee SF, Connolly S, Carignan A, Mazer CD, Loeb M, Mertz D. Prevention of Infections in Cardiac Surgery study (PICS): study protocol for a pragmatic cluster-randomized factorial crossover pilot trial. Trials. 2018 Dec 17;19(1):688. doi: 10.1186/s13063-018-3080-y. PMID 30558680